CLINICAL TRIAL: NCT03411083
Title: Silkeborg Knee Replacement Cohort Study
Status: Completed | Type: Observational
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 6500009
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2020-05

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Rehabilitation; Recovery of function; Outcome Assessment (Health Care); Patient Reported outcome Measures; Treatment Outcome; Pain, Postoperative; Pain Management; Orthopedic Surgery
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Knee replacement: Patients assigned for total or unicompartmental knee replacement surgery
  Interventions: Procedure: Total or unicompartmental knee replacement

INTERVENTIONS:
Procedure: Total or unicompartmental knee replacement — Fast-track Knee replacement surgery including same day surgery

SUMMARY:
In this cohort study, we will investigate short and long term outcomes after knee replacement surgery and identify preoperative and early postoperative factors associated with long term outcome.

DETAILED DESCRIPTION:
All patients follow the same fast-track program including same day surgery for elective knee replacement surgery at the Silkeborg Regional Hospital in Denmark, which includes detailed preoperative written information, multidisciplinary education course for patients and relatives, optimized multimodal pain treatment and early postoperative rehabilitation. Before the admission for surgery, patients will be asked to fulfill several questionnaires and baseline information regarding work situation, educational level and previous treatments. At two weeks there, there is a scheduled follow up by a physical therapist and a nurse at the hospital. At three months there is a scheduled follow up by telephone with a physical therapist.

The study will adhere methodologically to the STROBE guidelines and checklist for prospective cohort studies (www.strobe-statement.org).

Further description is provided elsewhere as eligibility criteria and outcome measures.

Addition to the description:

In January 2019 we started collecting 1 year follow-up data and included questions regarding treatment success, satisfaction and willingness to repeat the surgery.

In March 2019 we decided to make a change in the baseline collection of relevant predictors for primary outcome. The reason for the change was to be able to answer more relevant scientific questions in the cohort study. We replaced "The General Self-efficacy Scale" with "Pain Catastrophizing Scale" and excluded "The General Self-efficacy Scale" from the 12 weeks follow-up collection of outcome measures.

March 2020:

The SIKS study was planned to continue recruitment until reaching minimum 1,000 TKA patients with follow-up data which was deemed sufficient for the purpose of the planned studies. In March 2020, the COVID-19 pandemic closed down all elective orthopaedic surgeries. Because of that, we decided to stop the recruitment to the cohort study with the last patient included (at March 16th, 2020, prior to the COVID-19 lockdown).

December 2020:

The first substudies are planned using data from the SIKS cohort:

1. Predictors of knee pain and functional outcome following Total Knee Arthroplasty - a prospective cohort study with 12 months follow up

   Primary outcome:

   Oxford Knee Score at 12 months
2. Is it feasible and safe to discharge patients on the day of surgery after a total knee arthroplasty?

   Primary outcomes Feasibility measured as length of stay Safety measures as readmission (phone calls, outpatient visits and inpatient visits) and the related reason

   Secondary outcomes Oxfort knee score (90 days) Pain intensity (90 days)
3. Associations between preoperative BMI and postoperative physical activity level and functional capacity 12 months after UKA or TKA surgery.

   Primary outcome UCLA scale (12 months)

   Secondary outcomes Oxford Knee Score (12 months)

   February 2024
4. Opioid use at 3 and 12 months following primary knee arthroplasty: a prospective cohort study

Primary outcome: Patient-reported use of opioids 3 and 12 months after knee arthroplasty.

Secondary outcome: Patient-reported causes for opioid use 3 and 12 months after knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Assigned for primary Unicompartmental or Total Knee Replacement
* Age ≥ 18 years at the time of recruitment
* Able to read and understand Danish

Exclusion Criteria:

* Not mentally able to reply to the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients assigned for primary knee replacement in the period from February 2018 to May 2020 will be consecutively recruited to the cohort from Silkeborg Regional Hospital Denmark.
Sampling Method: Probability Sample
Enrollment: 1225 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Oxford Knee Score (OKS) (continous) | 52 weeks after surgery
  Disease specific Patient Reported Outcome Measure regarding function and pain. Each question is answered by ticking a box on a five-point Likert scale. Responses are then totalled to obtain a score between 0 and 48, with 48 being the best.

SECONDARY OUTCOMES:
Oxford Knee Score (OKS) (continous) | Pre surgery
  Disease specific Patient Reported Outcome Measure regarding function and pain. Each question is answered by ticking a box on a five-point Likert scale. Responses are then totalled to obtain a score between 0 and 48, with 48 being the best.
Oxford Knee Score (OKS) (continous) | 12 weeks after surgery
  Disease specific Patient Reported Outcome Measure regarding function and pain. Each question is answered by ticking a box on a five-point Likert scale. Responses are then totalled to obtain a score between 0 and 48, with 48 being the best
EQ-5D-5L (continous) | Pre surgery
  Generic Health Related Quality of Life Patient Reported Outcome Measure
EQ-5D-5L (continous) | 12 weeks after surgery
  Generic Health Related Quality of Life Patient Reported Outcome Measure
EQ-5D-5L (continous) | 52 weeks after surgery
  Generic Health Related Quality of Life Patient Reported Outcome Measure
The General Self-efficacy Scale (continous) | Pre surgery
  A generic Patient Reported Outcome Measure. The General Self-efficacy Scale measures self-efficacy, defined as an individual's belief in his or her capacity to execute behaviors necessary to produce specific performance attainments.Each question is answered by ticking a box on a four-point Likert scale. Responses are then totalled to obtain a score between 10 and 40, with 40 being the best. he General Self-efficacy Scale measures self-efficacy, defined as an individual's belief in his or her capacity to execute behaviors necessary to produce specific performance attainments.Each question is answered by ticking a box on a four-point Likert scale. Responses are then totalled to obtain a score between 10 and 40, with 40 being the best. The General Self-efficacy Scale is included in the data collection from January 2019 til March 2019, which corresponds to about 550 patient responds.
The General Self-efficacy Scale (continous) | 12 weeks after surgery
  A generic Patient Reported Outcome Measure. The General Self-efficacy Scale measures self-efficacy, defined as an individual's belief in his or her capacity to execute behaviors necessary to produce specific performance attainments. Each question is answered by ticking a box on a four-point Likert scale. Responses are then totalled to obtain a score between 10 and 40, with 40 being the best. The General Self-efficacy Scale is included in the data collection from January 2019 til June 2019, which corresponds to about 550 patient responds
Pain Visual Analog Scale (VAS) (continous) | Pre surgery
  Measured in rest and activity. The pain VAS is a generic pain measure on a continuous scale comprised of a horizontal line orientated from the left (worst) to the right (best), 100 mm in length
Pain Visual Analog Scale (VAS) (continous) | 12 weeks after surgery
  Measured in rest and activity. The pain VAS is a generic pain measure on a continuous scale comprised of a horizontal line orientated from the left (worst) to the right (best), 100 mm in length
Pain Visual Analog Scale (VAS) (continous) | 52 weeks after surgery
  Measured in rest and activity. The pain VAS is a generic pain measure on a continuous scale comprised of a horizontal line orientated from the left (worst) to the right (best), 100 mm in length
Analgetic pain medication intake (type and frequence) | Pre surgery
  Self-reported by the patients
Analgetic pain medication intake (type and frequence) | 12 weeks after surgery
  Self-reported by the patients
Analgetic pain medication intake (type and frequence) | 52 weeks after surgery
  Self-reported by the patients
Range of Motion (ROM) in passive knee flexion and passive knee extension (degrees) | Pre surgery
  Measures is conducted by a doctor
UCLA Activity Scale (continuous) | Pre surgery
  Patient Reported Outcome Measure, that measures physical activity in patients with knee replacements on a 10-level scale, where "10" is very active
UCLA Activity Scale (continuous) | 12 weeks after surgery
  Patient Reported Outcome Measure, that measures physical activity in patients with knee replacements on a 10-level scale, where "10" is very active
UCLA Activity Scale (continuous) | 52 weeks after surgery
  Patient Reported Outcome Measure, that measures physical activity in patients with knee replacements on a 10-level scale, where "10" is very active
Pain Catastrophizing Scale (PCS) | Pre surgery
  Patient Reported Outcome Measure, that measures how patients experience pain. Pain catastrophizing is characterized by the tendency to magnify the threat value of a pain stimulus and to feel helpless in the presence of pain, as well as by a relative inability to prevent or inhibit pain-related thoughts in anticipation of, during, or following a painful event such as surgery for example. Each of the 13 questions is answered by ticking a box on a 5 point Likert Scale from 0 (not at all) to 4 (all the time). A total score is yielded (ranging from 0-52 and 0 being the best), along with three subscale scores assessing rumination, magnification and helplessness. The PCS is included in the data collection from March 2019 til end of the cohort study, which corresponds to about 950 patient responses (instead of The General Self-efficacy Scale)
Global Perceived Effect (GPE) | 52 weeks after surgery
  GPE measures patients' perception of the change in their knee problems after the surgery. GPE will be assessed with the anchor question "Overall, how are the problems now (pain and ability to perform daily activities) in the knee on which you had surgery, compared to prior to your operation?" Patients respond on a 7-point scale ranging from "better, an important improvement" to "worse, an important deterioration".
Satisfaction with the surgery | 52 weeks after surgery
  Satisfaction is measured with the question "Overall, how satisfied are you with the sugery?". Patients respond on a 5 point scale ranging from "very satisfied" to "very unsatisfied"
Patient Acceptable Symptom State (PASS) | 52 weeks after surgery
  PASS measures satisfaction with the current knee function and will be assessed with the anchor question ""When you think of your knee function, will you consider your current condition as satisfying? With knee function, you should take into account your activities of daily living, your level of pain and other symptoms". Patients respond "yes" or "no". If patients respond "no" they are asked if the consider the treatment of ther knee problem as a failure.
Global assessment of willingness to repeat the surgery | 52 weeks after surgery
  Assessed with the anchor question "knowing what your knee arthroplasty surgery did for you, if you could go back in time, would you still have undergone this surgery?" Patients respond "yes", "no" or "uncertain".
Feasibility (length of stay) | 2 weeks after surgery
  Measured as length of stay and reason for not being discharged on post operative day 0 (same-day) will be provided.
Safety (readmission) | 1) 2 weeks after surgery, 2) 2 weeks after surgery, and 3) 90 days after discharge
  1. number of patient-initiated phone calls
  2. number of unscheduled visits in the outpatient clinic
  3. number of inpatient readmission (admission to hospital ward taking up a bed)
Safety (complications) | 1) 2 weeks after surgery, 2) 2 weeks after surgery, and 3) 90 days after discharge
  The reason for readmission (=complication) in relation to:
  1. patient-initiated phone calls
  2. unscheduled visits in the outpatient clinic
  3. inpatient readmission (admission to hospital ward taking up a bed) will be reported.

OTHER OUTCOMES:
Pain Visual Analog Scale (VAS) (continous) | 2 weeks after surgery
  Measured in rest and activity. The pain VAS is a generic pain measure on a continuous scale comprised of a horizontal line orientated from the left (worst) to the right (best), 100 mm in length
Analgetic pain medication intake (type and frequence) | 2 weeks after surgery
  Registrated by a nurse
Range of Motion (ROM) in passive knee flexion and passive knee extension (degrees) | 2 weeks after surgery
  Measures is conducted by a physical therapist
Range of Motion (ROM) in passive knee flexion and passive knee extension (degrees) | pre surgery
  Measures is conducted by a doctor

CONTACTS AND LOCATIONS:
Overall Officials: Lone Ramer Mikkelsen, Msc., Ph.D., Principal Investigator — Interdisciplinary Research Unit Elective Surgery Centre Silkeborg Regional Hospital, Denmark; Mette Garval, PT, Msc., Principal Investigator — Physical Therapy Department, Elective Surgery Centre Silkeborg Regional Hospital, Denmark; Søren Thorgaard Skou, PT, PhD, Study Chair — Research Unit for Musculoskeletal Function and Physiotherapy University of Southern Denmark; Anne Mette Schmidt, Msc., Ph.D., Principal Investigator — Interdisciplinary Research Unit Elective Surgery Centre Silkeborg Regional Hospital, Denmark
Locations (1):
- Silkeborg Regional Hospital, Silkeborg, Jutland, Denmark